CLINICAL TRIAL: NCT01541046
Title: Lactobacillus Reuteri DSM 17938 Versus Placebo in the Treatment of Infantile Colic: A Randomized Double-blind Controlled Trial
Brief Title: Lactobacillus Reuteri DSM 17938 Versus Placebo in the Treatment of Infantile Colic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Gideon Koren, Director of MotherRisk Program, Clinical Pharmacology and Toxicology, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000018504
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Colic
Keywords: pediatric; infantile colic; probiotic treatment
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biogaia L. reuteri DSM 17938 (Experimental): Biogaia L. reuteri DSM 17938, probiotic infant drops (5 drops=10^8 cfu),5 drops, once per day for 21 days.
  Interventions: Biological: Biogaia L. reuteri DSM 17938
- Probiotic Placebo (Placebo Comparator): Placebo drops (sunflower oil, medium chain triglyceride oil, silicon chloride), 5 drops, once a day for 21 days.
  Interventions: Biological: Probiotic Placebo

INTERVENTIONS:
Biological: Biogaia L. reuteri DSM 17938 — Freeze-dried Lactobacillus reuteri DSM 17938 suspended in oil. Brand Name Active Agent: BioGaia™
  Arms: Biogaia L. reuteri DSM 17938
Biological: Probiotic Placebo — Description of Placebo: contains same excipients as Active Agent, without the active ingredient
  Arms: Probiotic Placebo

SUMMARY:
Infantile colic is a common medical condition which remains a frustrating problem for parents and health care providers with no clear treatment guidelines. To fill the void in existing literature, we present a protocol to examine whether probiotics are effective in decreasing infantile colic symptoms when compared to placebo treatment.

We hypothesize that oral administration of the probiotic L. reuteri DSM 17938 will reduce symptoms of infantile colic in breastfed infants in comparison to placebo.

An interim analysis will be conducted after 50 infants randomized to monitor both safety and efficacy.

DETAILED DESCRIPTION:
Infantile colic is one of the most commonly reported medical problems within the first three months of life causing appreciable distress for both parents and pediatricians. The reported incidence of infantile colic ranges from 3% to 28% in prospective studies and up to 40% in retrospective surveys.

The pathogenesis of infantile colic remains elusive despite decades of research. It appears that multiple independent origins might be involved: amongst them infant's difficult temperament, inadequate mother-infant communication or maternal anxiety, transient lactase deficiency, exposure to cow's milk, abnormal gastrointestinal function, maternal smoking during pregnancy or after delivery. Consequently, various treatment approaches have been tried to alleviate this condition.

Recent studies have suggested that changes of intestinal microflora of a newborn may play an important role in pathogenesis of infantile colic. Therefore, dietary supplementation with probiotics has been proposed for the improvement of this condition.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy term infant 21-90 days of age
2. Birth weight ≥2500 g
3. Exclusively breastfed (to reduce variability in the intestinal microflora attributable to dietary variations)
4. With colic symptoms (>3 hours of crying on >3 days per week) with debut 10 ± 5 days before enrollment
5. Gestational age between 37 and 42 weeks
6. Apgar score higher than 7 at 5 minutes
7. Written informed consent from a parent

Exclusion Criteria:

1. Any chronic illness or gastrointestinal disorder as judged by the pediatrician
2. Any history of antibiotic treatment or probiotic supplementation
3. Failure to obtain a written consent by parent/legal guardian
4. Participation in other clinical trials
5. Infants with acute illness
6. Subjects with allergies or family history of allergies to any of the ingredients of the study product or placebo

Ages: 21 Days to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Mean change in crying time | Baseline, 7 days, 14 days, 21 days
  Reduction of daily median crying time (measured with parental diary) with L. reuteri DSM 17938 versus placebo at any of the time points 7, 14, and 21 days

SECONDARY OUTCOMES:
Number of responders vs. non-responders | Baseline, at 7, 14 and 21 days
  Number of responders versus non-responders with L. reuteri versus placebo at the time points 7, 14, and 21 days. Responder is defined as a decrease in daily average crying time of 50% during the study as measured using the maternal daily diary.
Parental quality of life | Daily for 21 days
  Parental quality of life assessed by self-administered numerical rating scale from 0 (worst possible) to 10 (perfect well-being)
Number of episodes of crying | Over 21 days
  Reduction in the number of episodes of crying (measured with parental diary) with L. reuteri DSM 17938 versus placebo
Duration of episodes of crying | Over 21 days
  Reduction in the duration of episodes of crying (measured with parental diary) with L. reuteri DSM 17938 versus placebo
Changes in stool consistency | Over 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Koren, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Chau K, Lau E, Greenberg S, Jacobson S, Yazdani-Brojeni P, Verma N, Koren G. Probiotics for infantile colic: a randomized, double-blind, placebo-controlled trial investigating Lactobacillus reuteri DSM 17938. J Pediatr. 2015 Jan;166(1):74-8. doi: 10.1016/j.jpeds.2014.09.020. Epub 2014 Oct 23. PMID 25444531